CLINICAL TRIAL: NCT01012817
Title: A Phase 1/2 Trial of ABT-888, an Inhibitor of Poly(ADP-ribose) Polymerase (PARP), and Topotecan (TPT) in Patients With Solid Tumors (Phase 1) and Relapsed Ovarian Cancer or Primary Peritoneal Cancer (Phase 2) After Prior Platinum Containing First-Line Chemotherapy
Brief Title: Veliparib and Topotecan Hydrochloride in Treating Patients With Solid Tumors, Relapsed or Refractory Ovarian Cancer, or Primary Peritoneal Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-00312; NCI-2011-00312 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 09-000742; MC0861; MAYO-MC0861; CDR0000657976; 8329 (Other: Mayo Clinic Cancer Center LAO); 8329 (Other: CTEP); P50CA136393 (NIH); U01CA069912 (NIH); UM1CA186686 (NIH)
Record Dates: First submitted 2009-11-11; First posted 2009-11-13 (Estimated); Results first posted 2023-07-19 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Malignant Solid Neoplasm; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Unresectable Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis; Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Pharmacogenomic Testing; Topotecan; veliparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (veliparib and topotecan hydrochloride) (Experimental): Patients receive veliparib PO on days 1-3, 8-10, and 15-17 (veliparib is omitted on days 1-3 of course 2) and topotecan hydrochloride IV over 30 minutes on days 2, 9, and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Pharmacogenomic Study; Other: Pharmacological Study; Drug: Topotecan Hydrochloride; Drug: Veliparib

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacogenomic Study — Correlative studies
  Other Names: PHARMACOGENOMIC
Other: Pharmacological Study — Correlative studies
Drug: Topotecan Hydrochloride — Given IV
  Other Names: Evotopin; Hycamptamine; Hycamtin; Nogitecan Hydrochloride; Potactasol; SKF S 104864 A; SKF S-104864-A; SKF S104864A; Topotec; Topotecan HCl; topotecan hydrochloride (oral)
Drug: Veliparib — Given PO
  Other Names: ABT 888; ABT-888; ABT888; PARP-1 inhibitor ABT-888

SUMMARY:
This phase I/II trial studies the side effects and best dose of veliparib and topotecan hydrochloride and to see how well they work in treating patients with solid tumors, ovarian cancer that has come back or does not respond to treatment, or primary peritoneal cancer. Veliparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as topotecan hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving veliparib with chemotherapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose of the combination of veliparib (ABT-888) and weekly topotecan (topotecan hydrochloride) in adult patients with advanced solid tumors. (Phase I) II. To identify any anti-tumor activity of this treatment combination, as assessed by objective response in patients with advanced solid tumors. (Phase I) III. To assess the confirmed response rate for patients with epithelial ovarian cancer, fallopian tube cancer or primary peritoneal carcinoma treated with the combination of ABT-888 and weekly topotecan.

IV. To assess the progression free response (PFS) for patients with epithelial ovarian cancer, fallopian tube cancer or primary peritoneal carcinoma treated with the combination of ABT-888 and weekly topotecan. (Phase II)

SECONDARY OBJECTIVES:

I. To identify any pharmacokinetic interactions between ABT-888 and topotecan. (Phase I) II. To determine whether topotecan stimulates adenosine diphosphate (ADP)-ribose polymer formation in circulating peripheral blood mononuclear cells. (Phase I) III. To determine whether ABT-888 inhibits basal or topotecan-stimulated ADP-ribose polymer formation. (Phase I) IV. To assess differences in the toxicity and/or efficacy of this regimen based on BRCA 1/2 mutational status. (Phase II) V. To determine whether pretreatment tumor cell levels of topoisomerase I, poly ADP-ribose polymerase (PARP), BRCA1, BRCA2, XRCC1, tyrosyl-deoxyribonucleic acid (DNA) phosphodiesterase 1 (TDP1), P-glycoprotein or breast cancer resistance protein (BCRP) predict response to this regimen. (Phase II) VI. To identify, in an exploratory manner, any transcriptional profiles that may predict response to this regimen. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of veliparib and topotecan hydrochloride followed by a phase II study. (PHASE I DOSE-ESCALATION PART IS COMPLETED)

Patients receive veliparib orally (PO) on days 1-3, 8-10, and 15-17 (veliparib is omitted on days 1-3 of course 2) and topotecan hydrochloride intravenously (IV) over 30 minutes on days 2, 9, and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 3 months (Phase I) or every 3 or 6 months for 5 years (Phase II).

ELIGIBILITY:
Inclusion Criteria:

* PHASE I: Adult patients with histologically confirmed solid tumor malignancy that is metastatic or unresectable and for which standard curative measures or other therapy definitely capable of extending life expectancy does not exist
* PHASE II: All patients enrolled in the Phase II portion of this trial must have a history of biopsy-proven ovarian, fallopian tube or primary peritoneal cancer
* Patients must have received < 3 lines of prior therapy and have relapsed less than a year from their last platinum regimen; regimens that are used twice (for example carboplatin and paclitaxel) can be counted as one; if a regimen is changed during the course of treatment due to side effect profile or allergy, the course of therapy is counted as one regimen; (for example, if docetaxel is substituted for paclitaxel due to a reaction during the initial course of adjuvant therapy, this is considered one regimen)
* Patients must have measurable disease with at least one lesion whose longest diameter can be accurately measured as >= 2.0 cm with conventional techniques or as >= 1.0 cm with spiral computed topography (CT); if spiral CT is used, it must be used for both pre- and post- treatment tumor assessments
* Absolute neutrophil count >= 1500/mcL
* Hemoglobin >= 9.0 g/dL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x the upper limit of normal (ULN)
* Serum glutamic pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) or serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 2.5 x ULN in the absence of hepatic metastasis; SGPT (ALT) =< 3 x ULN or SGOT (AST) =< 5 x ULN in the presences of hepatic metastasis
* Creatinine =< 1.5 x ULN
* International normalized ratio (INR) =< 1.4 unless receiving therapeutic doses of coumadin
* Partial thromboplastin time (PTT) =< 48 seconds (1.25 x ULN)
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Ability to provide informed consent
* Willingness to return to enrolling institution for follow up
* Life expectancy >= 12 weeks
* Willingness to provide the biologic specimens is required by the protocol; this is part of the mandatory correlative research component; these specimens include:

  * PHASE I: peripheral blood for plasma pharmacokinetic analysis and peripheral blood mononuclear cell (PBMC) polymer assessment from 0-24 h after drug administration on days 1 and 2 of cycle 1 as well as day 2 of cycle 2; urine for assessment of ABT-888 renal clearance for 24 h after administration of drugs on days 1 and 2 of cycle 1 as well as day 2 of cycle 2; and a pretreatment peripheral blood sample for possible sequencing of the BRCA1, BRCA2 loci as well as possible pharmacogenomic analysis
* Negative urine or serum pregnancy test done =< 7 days prior to registration for females of child bearing potential only
* Able to swallow and absorb the medication

Exclusion Criteria:

* Known standard therapy for the patient's disease that is potentially curative or definitely capable of extending life expectancy
* Prior treatment with a PARP inhibitor or topotecan
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Any of the following prior therapies:

  * Chemotherapy =< 4 weeks prior to registration
  * Mitomycin C/nitrosoureas =< 6 weeks prior to registration
  * Immunotherapy =< 4 weeks prior to registration
  * Biologic therapy =< 4 weeks prior to registration
  * Radiation therapy =< 4 weeks prior to registration
  * Radiation to > 25% of bone marrow
  * Investigational therapy or any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation) =< 4 weeks prior to registration; subjects with prostate cancer will be permitted to continue hormone therapy
* Failure to fully recover from acute, reversible effects of prior chemotherapy regardless of interval since last treatment
* New York Heart Association classification III or IV
* Known central nervous system (CNS) metastases or seizure disorder; patients with known brain metastases that have been successfully treated and stable for >= 6 months without requirement for corticosteroids and without seizure activity will be eligible
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients (other than that related to the use of corticosteroids) including patients known to be human immunodeficiency virus (HIV) positive
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy, except non-melanotic skin cancer or carcinoma-in-situ of the cervix

  * Note: If there is a history of prior malignancy, they must not be receiving other specific treatment (other than hormonal therapy) for their cancer
* History of myocardial infarction =< 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* More than 2 prior chemotherapy regimens for the current malignancy; full dose chemotherapy used in conjunction with concurrent radiation therapy will be included as prior therapy

  * Note: Prior hormonal therapy (e.g. leuprolide, aromatase inhibitors, tamoxifen) and immunotherapy will be allowed and not included as a prior chemotherapy; if the chemotherapy regimen is altered during the course due to issues with tolerability or safety, the regimen will be counted as one; using the same regimen at recurrence is counted as one regimen; the addition of bevacizumab to a prior regimen is considered one regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2009-11-03 (Actual); Primary Completion 2019-01-13 (Actual); Study Completion 2026-08-27 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea E Wahner Hendrickson, Principal Investigator — Mayo Clinic Cancer Center LAO
Locations (15):
- United States (15):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 Dose Level 1: Patients receive 10qd veliparib PO on days 1-3, 8-10, and 15-17 (veliparib is omitted on days 1-3 of course 2) and 2mg/m^2 topotecan hydrochloride IV over 30 minutes on days 2, 9, and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Phase 1 Dose Level 2: Patients receive 20qd veliparib PO on days 1-3, 8-10, and 15-17 (veliparib is omitted on days 1-3 of course 2) and 2mg/m^2 topotecan hydrochloride IV over 30 minutes on days 2, 9, and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Phase 1 Dose Level 3: Patients receive 10qd veliparib PO on days 1-3, 8-10, and 15-17 (veliparib is omitted on days 1-3 of course 2) and 3mg/m^2 topotecan hydrochloride IV over 30 minutes on days 2, 9, and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Phase 1 Dose Level 4: Patients receive 20qd veliparib PO on days 1-3, 8-10, and 15-17 (veliparib is omitted on days 1-3 of course 2) and 3mg/m^2 topotecan hydrochloride IV over 30 minutes on days 2, 9, and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Phase 1 Dose Level 5: Patients receive 20qd veliparib PO on days 1-3, 8-10, and 15-17 (veliparib is omitted on days 1-3 of course 2) and 4mg/m^2 topotecan hydrochloride IV over 30 minutes on days 2, 9, and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Phase 1 Dose Level 6: Patients receive 30qd veliparib PO on days 1-3, 8-10, and 15-17 (veliparib is omitted on days 1-3 of course 2) and 4mg/m^2 topotecan hydrochloride IV over 30 minutes on days 2, 9, and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Phase 1 Dose Level 7: Patients receive 30qd veliparib PO on days 1-3, 8-10, and 15-17 (veliparib is omitted on days 1-3 of course 2) and 3mg/m^2 topotecan hydrochloride IV over 30 minutes on days 2, 9, and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Phase 1 Dose Level 8: Patients receive 50qd veliparib PO on days 1-3, 8-10, and 15-17 (veliparib is omitted on days 1-3 of course 2) and 3mg/m^2 topotecan hydrochloride IV over 30 minutes on days 2, 9, and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Phase 1 Dose Level 9: Patients receive 100qd veliparib PO on days 1-3, 8-10, and 15-17 (veliparib is omitted on days 1-3 of course 2) and 3mg/m^2 topotecan hydrochloride IV over 30 minutes on days 2, 9, and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Phase 1 Dose Level 10: Patients receive 150qd veliparib PO on days 1-3, 8-10, and 15-17 (veliparib is omitted on days 1-3 of course 2) and 3mg/m^2 topotecan hydrochloride IV over 30 minutes on days 2, 9, and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Phase 1 Dose Level 11: Patients receive 200qd veliparib PO on days 1-3, 8-10, and 15-17 (veliparib is omitted on days 1-3 of course 2) and 3mg/m^2 topotecan hydrochloride IV over 30 minutes on days 2, 9, and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Phase 1 Dose Level 12; Phase 2: Patients receive 300qd veliparib PO on days 1-3, 8-10, and 15-17 (veliparib is omitted on days 1-3 of course 2) and 3mg/m^2 topotecan hydrochloride IV over 30 minutes on days 2, 9, and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Phase 1 Dose Level 13: Patients receive 400qd veliparib PO on days 1-3, 8-10, and 15-17 (veliparib is omitted on days 1-3 of course 2) and 3mg/m^2 topotecan hydrochloride IV over 30 minutes on days 2, 9, and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 1 Dose Level 3 | Phase 1 Dose Level 4 | Phase 1 Dose Level 5 | Phase 1 Dose Level 6 | Phase 1 Dose Level 7 | Phase 1 Dose Level 8 | Phase 1 Dose Level 9 | Phase 1 Dose Level 10 | Phase 1 Dose Level 11 | Phase 1 Dose Level 12 | Phase 1 Dose Level 13 | Phase 2
Started | 3 | 3 | 3 | 4 | 6 | 7 | 3 | 4 | 3 | 6 | 5 | 7 | 3 | 31
Completed | 3 | 3 | 3 | 3 | 6 | 6 | 3 | 3 | 3 | 6 | 3 | 6 | 3 | 29
Not Completed | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 1 Dose Level 3 | Phase 1 Dose Level 4 | Phase 1 Dose Level 5 | Phase 1 Dose Level 6 | Phase 1 Dose Level 7 | Phase 1 Dose Level 8 | Phase 1 Dose Level 9 | Phase 1 Dose Level 10 | Phase 1 Dose Level 11 | Phase 1 Dose Level 12 | Phase 1 Dose Level 13 | Phase 2 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 6 | 7 | 3 | 4 | 3 | 6 | 5 | 7 | 3 | 31 | 88
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 52 [47 to 56] | 58.7 [53 to 64] | 67.7 [59 to 77] | 62.3 [51.5 to 73] | 60.3 [57 to 64] | 59.7 [52 to 70] | 50.3 [45 to 59] | 52 [50 to 54] | 54 [46 to 66] | 56.2 [49 to 64] | 56.2 [56 to 57] | 50.1 [41 to 65] | 55 [50 to 63] | 60.8 [53 to 69] | 58.0 [50 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 4 | 6 | 6 | 3 | 4 | 3 | 6 | 5 | 7 | 3 | 31 | 87
  Male | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3
  Not Hispanic or Latino | 3 | 3 | 3 | 4 | 6 | 7 | 3 | 4 | 3 | 6 | 5 | 6 | 2 | 29 | 84
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 3 | 3 | 6 | 6 | 3 | 4 | 3 | 6 | 4 | 7 | 2 | 30 | 83
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Topotecan Hydrochloride and Veliparib, Determined According to Incidence of Dose-limiting Toxicity, Graded Using National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (Phase I)
Description: The number of patients with a dose limiting toxicity will be reported. Dose-limiting toxicity (DLT) will be defined as a cycle 1 adverse event attributed (definitely, probably, or possibly) to the study treatment and meeting the following criteria: Grade 4 anemia, grade 4 neutrophil count decrease, grade 4 platelet count decrease, Serum creatinine >= 2 times baseline or ≥ 2 times the upper limit of normal if baseline is < the upper limit of normal, or other >= Grade 3 as per NCI Common Terminology Criteria for Adverse Events CTCAE version 4.0. >= Grade 3 nausea, vomiting, or diarrhea with maximal supportive treatment(s) will be considered dose-limiting. Grade 3 fatigue or anorexia will not be considered dos
Time Frame: 4 weeks
Population: All phase 1 patients that received treatment per protocol and evaluated for adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 1 Dose Level 3 | Phase 1 Dose Level 4 | Phase 1 Dose Level 5 | Phase 1 Dose Level 6 | Phase 1 Dose Level 7 | Phase 1 Dose Level 8 | Phase 1 Dose Level 9 | Phase 1 Dose Level 10 | Phase 1 Dose Level 11 | Phase 1 Dose Level 12 | Phase 1 Dose Level 13
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 3 | 3 | 3 | 6 | 3 | 6 | 3
Participants | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 2

2. Primary Outcome: Percent of Patients With Tumor Response, Defined as Complete Response or Partial Response as Assessed Using Response Evaluation Criteria In Solid Tumors
Description: The proportion of successes will be estimated by the number of successes(CR or PR) divided by the total number of evaluable patients. Confidence intervals for the true success proportion will be calculated according to the approach of Duffy and Santner (1987). Complete Response (CR) is defined as disappearance of all target lesions and, if non target lesions exist, the disappearance of all non-target lesions and normalization of tumor maker level. At least 30% decrease in the sum of the longest diameter (LD) of target lesion taking as reference the baseline sum.
Time Frame: Up to 48 weeks (12 courses)
Population: All treated patients that were evaluated for disease response
Measure: Number; unit: percent of patients with response
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 1 Dose Level 3 | Phase 1 Dose Level 4 | Phase 1 Dose Level 5 | Phase 1 Dose Level 6 | Phase 1 Dose Level 7 | Phase 1 Dose Level 8 | Phase 1 Dose Level 9 | Phase 1 Dose Level 10 | Phase 1 Dose Level 11 | Phase 1 Dose Level 12 | Phase 1 Dose Level 13 | Phase 2
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 3 | 3 | 3 | 6 | 3 | 6 | 3 | 29
percent of patients with response | 0 | 33 | 0 | 0 | 17 | 0 | 0 | 0 | 0 | 0 | 0 | 50 | 0 | 0

3. Secondary Outcome: Overall Survival
Description: The distribution of survival time for phase 2 patients will be estimated using the method of Kaplan-Meier.
Time Frame: The time from registration to death due to any cause, assessed up to 5 years
Reporting Status: Not Posted, anticipated posting 2026-08

4. Secondary Outcome: Progression Free Survival
Description: The distribution of progression free survival will be estimated using the method of Kaplan-Meier.
Time Frame: The time from registration to the earliest date of documentation of disease progression or death due to any cause, assessed up to 5 years
Reporting Status: Not Posted, anticipated posting 2026-08

5. Secondary Outcome: Duration of Response
Description: Duration of response is defined for all evaluable patients who have achieved an objective response as the date at which the patient's earliest best objective status is first noted to be either a complete response or partial response to the earliest date progression is documented.
Time Frame: Up to 5 years
Reporting Status: Not Posted, anticipated posting 2026-08

6. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure is defined to be the time from the date of registration to the date at which the patient is removed from treatment due to progression, adverse events, or refusal.
Time Frame: The time from the date of registration to the date at which the patient is removed from treatment due to progression, adverse events, or refusal, assessed up to 5 years
Reporting Status: Not Posted, anticipated posting 2026-08

7. Secondary Outcome: Adverse Events, Graded Using National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0
Description: The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 75 months
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 10 | Phase 1 Dose Level 11 | Phase 1 Dose Level 12 | Phase 1 Dose Level 13 | Phase 2 | Phase 1 Dose Level 2 | Phase 1 Dose Level 3 | Phase 1 Dose Level 4 | Phase 1 Dose Level 5 | Phase 1 Dose Level 6 | Phase 1 Dose Level 7 | Phase 1 Dose Level 8 | Phase 1 Dose Level 9
All-Cause Mortality (participants affected / at risk) | 0/3 | 2/6 | 0/5 | 1/7 | 1/3 | 2/31 | 0/3 | 1/3 | 1/4 | 1/6 | 1/7 | 1/3 | 0/4 | 1/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/6 | 3/5 | 5/7 | 2/3 | 12/31 | 0/3 | 1/3 | 1/4 | 3/6 | 2/7 | 2/3 | 1/4 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 5/5 | 7/7 | 3/3 | 29/31 | 3/3 | 3/3 | 4/4 | 6/6 | 7/7 | 3/3 | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Level 1 (N=3) | Phase 1 Dose Level 10 (N=6) | Phase 1 Dose Level 11 (N=5) | Phase 1 Dose Level 12 (N=7) | Phase 1 Dose Level 13 (N=3) | Phase 2 (N=31) | Phase 1 Dose Level 2 (N=3) | Phase 1 Dose Level 3 (N=3) | Phase 1 Dose Level 4 (N=4) | Phase 1 Dose Level 5 (N=6) | Phase 1 Dose Level 6 (N=7) | Phase 1 Dose Level 7 (N=3) | Phase 1 Dose Level 8 (N=4) | Phase 1 Dose Level 9 (N=3)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ECG QT corrected interval prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Oth spec (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Dose Level 1 (N=3) | Phase 1 Dose Level 10 (N=6) | Phase 1 Dose Level 11 (N=5) | Phase 1 Dose Level 12 (N=7) | Phase 1 Dose Level 13 (N=3) | Phase 2 (N=31) | Phase 1 Dose Level 2 (N=3) | Phase 1 Dose Level 3 (N=3) | Phase 1 Dose Level 4 (N=4) | Phase 1 Dose Level 5 (N=6) | Phase 1 Dose Level 6 (N=7) | Phase 1 Dose Level 7 (N=3) | Phase 1 Dose Level 8 (N=4) | Phase 1 Dose Level 9 (N=3)
Anemia (Blood and lymphatic system disorders) | 3 (40) | 6 (36) | 5 (22) | 6 (53) | 3 (21) | 21 (45) | 2 (5) | 3 (5) | 4 (11) | 6 (112) | 4 (34) | 2 (6) | 3 (33) | 1 (5)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 0 (0) | 4 (15) | 2 (7) | 0 (0) | 1 (1) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (18) | 1 (2) | 1 (4) | 3 (12) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (4) | 1 (1) | 1 (2) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (4) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (11) | 3 (4) | 4 (6) | 3 (20) | 1 (5) | 8 (17) | 2 (9) | 1 (3) | 2 (3) | 5 (20) | 2 (6) | 2 (4) | 2 (3) | 1 (2)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (2) | 1 (6) | 0 (0) | 0 (0) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bloating (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 2 (3) | 1 (8) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (2)
Colonic hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Colonic obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (10) | 3 (12) | 2 (8) | 3 (10) | 2 (5) | 12 (25) | 2 (8) | 2 (2) | 2 (2) | 3 (7) | 1 (5) | 2 (4) | 4 (8) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (5) | 3 (12) | 3 (6) | 5 (20) | 3 (7) | 8 (18) | 1 (8) | 0 (0) | 4 (5) | 3 (39) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (13) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (15) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (8) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 0 (0) | 2 (4) | 2 (14) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 1 (3) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (11) | 0 (0) | 1 (3) | 1 (7) | 0 (0) | 0 (0) | 3 (8) | 1 (4) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (21) | 5 (24) | 5 (10) | 6 (32) | 3 (9) | 19 (48) | 2 (10) | 1 (1) | 3 (8) | 6 (71) | 5 (13) | 2 (11) | 4 (16) | 2 (5)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 5 (18) | 3 (3) | 6 (21) | 3 (10) | 13 (25) | 1 (2) | 0 (0) | 4 (11) | 4 (29) | 4 (5) | 1 (5) | 3 (11) | 2 (2)
Chills (General disorders) | 1 (2) | 1 (1) | 2 (2) | 4 (13) | 1 (2) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 3 (12) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 2 (3) | 1 (1) | 2 (9) | 0 (0) | 3 (6) | 0 (0) | 1 (1) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (27) | 6 (17) | 3 (6) | 6 (33) | 3 (9) | 16 (50) | 2 (9) | 2 (5) | 2 (3) | 5 (50) | 4 (12) | 2 (12) | 2 (3) | 1 (2)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (8) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (5) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (8)
Gen disord and admin site conds-Oth spec (General disorders) | 0 (0) | 2 (9) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck edema (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 2 (7) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (10) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (8) | 1 (3) | 0 (0) | 1 (7) | 0 (0) | 5 (10) | 0 (0) | 1 (1) | 0 (0) | 2 (7) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune system disorders - Other, specify (Immune system disorders) | 0 (0) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infections and infestations - Oth spec (Infections and infestations) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 1 (2) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (17) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial throm time prolonged (Investigations) | 0 (0) | 2 (3) | 2 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (19) | 3 (7) | 0 (0) | 2 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 3 (5) | 1 (1) | 1 (3) | 0 (0) | 4 (4) | 1 (2) | 1 (2) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (1) | 0 (0) | 1 (2) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 2 (4) | 0 (0) | 2 (13) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ECG QT corrected interval prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INR increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (8) | 1 (10) | 0 (0) | 1 (14) | 0 (0)
Investigations - Other, specify (Investigations) | 1 (3) | 0 (0) | 2 (2) | 2 (5) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 5 (40) | 2 (4) | 1 (3) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 2 (6) | 2 (5) | 3 (9) | 3 (16) | 1 (8) | 7 (17) | 0 (0) | 0 (0) | 1 (1) | 3 (10) | 2 (4) | 1 (9) | 2 (9) | 1 (3)
Lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (16) | 6 (23) | 3 (16) | 5 (32) | 2 (8) | 15 (31) | 2 (11) | 2 (3) | 3 (10) | 6 (41) | 6 (32) | 1 (3) | 2 (8) | 1 (5)
Platelet count decreased (Investigations) | 1 (19) | 6 (21) | 3 (13) | 5 (15) | 2 (6) | 20 (44) | 2 (6) | 2 (2) | 2 (6) | 5 (87) | 5 (34) | 1 (1) | 2 (9) | 1 (1)
Weight loss (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
White blood cell decreased (Investigations) | 1 (32) | 6 (29) | 4 (26) | 5 (38) | 3 (9) | 14 (37) | 2 (9) | 2 (2) | 2 (7) | 4 (44) | 5 (29) | 1 (13) | 3 (23) | 1 (5)
Anorexia (Metabolism and nutrition disorders) | 2 (5) | 5 (18) | 3 (4) | 5 (20) | 3 (7) | 7 (11) | 1 (7) | 2 (4) | 3 (7) | 3 (30) | 3 (6) | 2 (10) | 2 (3) | 2 (10)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 4 (7) | 3 (3) | 2 (6) | 2 (2) | 4 (15) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3) | 1 (2) | 3 (5) | 1 (4) | 3 (7) | 2 (5) | 1 (1) | 2 (2) | 2 (4) | 3 (4) | 3 (7) | 0 (0) | 1 (3) | 1 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (6) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (33) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 2 (6) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 2 (3) | 1 (5) | 1 (1) | 1 (3) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (15) | 0 (0) | 1 (1) | 0 (0) | 2 (5) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (26) | 1 (4) | 1 (1) | 1 (3) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (5) | 0 (0) | 3 (8) | 2 (3) | 0 (0) | 1 (2) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 1 (1) | 2 (8) | 1 (1) | 2 (12) | 1 (1) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (11) | 3 (7) | 1 (1) | 3 (9) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 2 (4) | 1 (4) | 0 (0) | 1 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (6) | 0 (0) | 0 (0) | 1 (23) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (22) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (8) | 0 (0) | 0 (0) | 1 (8) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (7) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (14) | 1 (2) | 1 (5) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (11) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concentration impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 1 (1) | 2 (7) | 1 (2) | 1 (4) | 1 (7) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Dysphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 3 (8) | 3 (16) | 1 (2) | 1 (7) | 3 (5) | 7 (12) | 1 (9) | 1 (1) | 1 (1) | 5 (42) | 2 (3) | 1 (3) | 1 (10) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervous system disorders - Oth spec (Nervous system disorders) | 0 (0) | 1 (11) | 0 (0) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (4) | 1 (1) | 1 (1) | 2 (11) | 0 (0) | 4 (13) | 1 (8) | 0 (0) | 1 (2) | 2 (16) | 0 (0) | 1 (6) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (9) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (7) | 1 (2) | 2 (2) | 3 (9) | 1 (3) | 5 (15) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (6) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 4 (18) | 0 (0) | 0 (0) | 0 (0) | 1 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (2) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (15) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (19) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 0 (0) | 1 (2) | 2 (4) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (36) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (6) | 0 (0) | 4 (6) | 0 (0) | 2 (2) | 1 (2) | 1 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (7) | 0 (0) | 4 (6) | 0 (0) | 7 (17) | 1 (7) | 1 (3) | 0 (0) | 4 (48) | 1 (2) | 2 (6) | 1 (2) | 1 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (7) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 3 (9) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (17) | 2 (10) | 1 (4) | 2 (17) | 3 (7) | 6 (25) | 1 (2) | 0 (0) | 1 (1) | 4 (45) | 4 (10) | 1 (11) | 1 (10) | 1 (10)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (8) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (19) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 5 (11) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 0 (0) | 2 (3) | 3 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (7) | 0 (0) | 4 (7) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Superficial thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-13): https://cdn.clinicaltrials.gov/large-docs/17/NCT01012817/Prot_SAP_000.pdf